CLINICAL TRIAL: NCT00240695
Title: An Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of Galantamine HBr in the Treatment of Mild Cognitive Impairment
Brief Title: A Follow-up Study to Assess Safety and Tolerability of Galantamine Treatment in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005947
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Cognition Disorder; Nervous System Diseases; Mental Disorders; Brain Diseases
Keywords: Alzheimer's disease; Dementia; Brain Disease; Memory Loss; galantamine; Nervous System Diseases; open-label; elderly
MeSH Terms: conditions — Cognition Disorders; Nervous System Diseases; Mental Disorders; Brain Diseases; Alzheimer Disease; Dementia; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this follow-up study is to assess the long-term safety and tolerability of galantamine in individuals with mild cognitive impairment who participated in a previous study with galantamine

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose ability to perform daily tasks related to personal care (for example bathing, dressing, eating) and may be unable to handle money or travel to familiar places. The term mild cognitive impairment (MCI) is used to describe individuals who have memory impairments suggestive of early dementia, but do not yet meet the criteria for Alzheimer's disease. Individuals with MCI are more likely to develop Alzheimer's disease than normal elderly patients. Individuals with MCI who completed 1 of 2 previous double-blind studies with galantamine may participate in this follow-up study if they have not progressed to dementia. They will receive open-label galantamine for 12 months and will be evaluated after 2, 6 and 12 months of treatment. Safety evaluations (incidence of adverse events, ECGs, physical examinations, laboratory tests) will be performed throughout the study. Effectiveness will be assessed after 12 months of treatment (by using standardized tests and rating scales (Alzheimer's Disease Assessment Scale: cognitive/MCI version [ADAS-Cog/MCI], Clinical Dementia Rating [CDR] and CDR-Sum of the Boxes [CDR-SB]). Health status will be assessed using the Health Survey portion of the Short-Form 36 (SF-36) and the use of health and social care resources will be assessed using a resource-use questionnaire. The enrolled individuals may participate in an optional portion of the study in which their genetic material is analyzed to see if contains something that would affect the way galantamine is used by their bodies. Galantamine 8 or 12 milligrams (mg) by mouth twice daily for 12 months. Dose will start at 4 mg twice daily and be gradually increased to final dose; 12 mg twice daily dose may be decreased to 8 mg twice daily based upon tolerability

ELIGIBILITY:
Inclusion Criteria:

* Completed 24 months of double-blind treatment in 1 of 2 previous studies with galantamine without progressing to dementia (CDR< 1)
* Able to safely receive open-label galantamine in the opinion of the investigator and treatment is in the individual's best interest
* Regular (at least 3 days a week) visits from a person able to accompany patient to scheduled visits
* Enrolled within 7-30 days after the previous galantamine study Exclusion Criteria:
* Individuals who converted to dementia (CDR > = 1) during 1 of the previous galantamine studies
* Prematurely discontinued 1 of the previous galantamine studies or completed 1 of the previous studies more than 30 days prior to this study
* Current clinically significant cardiovascular disease (including heart surgery, unstable angina, congestive heart failure, fibrillation, valve disease or uncontrolled high blood pressure)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2003-05; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events; Changes in laboratory tests, ECGs, and physical examinations

SECONDARY OUTCOMES:
Change in CDR, ADAS-Cog/MCI version, CDR-SB and SF-36 scores from baseline to end of treatment; resource use; time to conversion to dementia

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A follow-up study to assess safety and tolerability of galantamine treatment in patients with mild cognitive impairment — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=688&filename=CR005947_CSR.pdf